CLINICAL TRIAL: NCT07375771
Title: Interventional Study to Evaluate the Effectiveness of Transcranial Alternating Current Stimulation (tACS) on Cognitive Performance in Patients With Lewy Body Dementia
Brief Title: Transcranial Alternating Current Stimulation in Lewy Body Dementia
Acronym: TACSDLB2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Responsible Party: Principal Investigator, Prof. Barbara Borroni, Professor, IRCCS Centro San Giovanni di Dio Fatebenefratelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TACSDLB2
Record Dates: First submitted 2025-12-01; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-09

CONDITIONS: Lewy Body Dementia (LBD); Transcranial Alternating Current Stimulation
MeSH Terms: conditions — Lewy Body Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The study is a double-blind, randomised and placebo-controlled trial, participants will be randomised into two groups: group 1, participants will receive real tACS for 2 weeks; and group 2, placebo tACS 2 weeks.
  Each participant will receive a total of 2 weeks of intervention, with 5 sessions per week (Wednesday to Tuesday) lasting approximately 60 minutes each.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Real tACS (Experimental): 10 sessions of Transcranial Alternating Current Stimulation (5 sessions/week, 60 minutes/session)
  Interventions: Device: Transcranial Alternating Current Stimulation
- Sham Comparator: Sham tACS (Sham Comparator): 10 sessions of sham Transcranial Alternating Current Stimulation (5 sessions/week, 60 minutes/session)
  Interventions: Device: Sham Transcranial Alternating Current Stimulation

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation — 10 sessions (5 days/week for 2 weeks), each consisting in the application of a tACS session (real at 3 mA) at the cortical level for a duration of 60 minutes each.
  Arms: Experimental: Real tACS
Device: Sham Transcranial Alternating Current Stimulation — 10 sessions (5 days/week for 2 weeks), each consisting in the application of a sham tACS session at the cortical level for a duration of 60 minutes each. The electrode placement will be identical to that used for real stimulation. However, the electrical current will be automatically interrupted approximately 5 seconds after the start of stimulation, making it impossible for the patient to distinguish between sham and real stimulation
  Arms: Sham Comparator: Sham tACS

SUMMARY:
The aim of the study is to evaluate the safety, feasibility, clinical and biological efficacy, and predictors of efficacy of an intervention consisting of transcranial alternating current stimulation (tACS) in patients with Lewy Body Dementia (DLB).

In neurodegenerative diseases, like DLB, the process of neurodegeneration is accompanied by a significant alteration in oscillatory activity.

tACS is a neurophysiological method of non-invasive modulation of the excitability of the central nervous system that uses a mild electrical current. Recent studies have demonstrated the safety and efficacy of this method in modulating the natural brain oscillation frequencies underlying multiple cognitive processes, such as verbal memory, perception, and working memory. Preliminary data show that single stimulation with occipital α-tACS results in a significant improvement in visuospatial abilities and executive functions in patients wih DLB.

The study is double blind, randomised and placebo-controlled, participants will be randomised into two groups: group 1, participants will receive real tACS for 2 weeks, from Wednesday to Tuesday (5 sessions/week, lasting approximately 60 minutes each); and group 2, participants will receive placebo tACS for 2 weeks (5 sessions/week, lasting approximately 60 minutes each).

Visits will take place at the beginning of the study (T00), after 2 weeks (T02), and 12 weeks (T12, follow-up). During each visit, participants undergo the following procedures: (i) blood sampling, (ii) clinical and neuropsychological assessment, (iii) EEG, and (iv) TMS-EEG. The occurrence of adverse events will be monitored throughout the duration of the study. Specific biomarker analyses will be performed on the blood samples to study the pathophysiological mechanisms of the disease and the effect of the experimental intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged over 18 at the time of signing the informed consent form;
* Presence of a clinical diagnosis of Lewy body dementia according to clinical criteria (McKeith et al., 2017)

Exclusion Criteria:

* Age younger than that stated in the inclusion criteria;
* Incapacity to understand;
* Contraindications for tACS and TMS: patients with cardiac pacemakers and metal implants that are not compatible with electric or magnetic fields, history of epilepsy, current pregnancy (Safety questionnaire)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events of Transcranial Alternating Current Stimulation Protocol | Through study completion, at week 12
  Safety and tolerability will be assessed in terms of incidence and severity of any adverse events. Safety and tolerability will be monitored throughout the duration of the study.
Feasibility of Transcranial Alternating Current Stimulation Protocol | Through study completion, at week 12
  Feasibility will be assessed based on the drop-out rate. Feasibility will be monitored throughout the duration of the study.
Mini-Mental State Examination (MMSE) | Change from baseline to week 12
  The global cognitive functioning will be assessed by Mini-Mental State Examination (MMSE); MMSE scores range from 0 to 30, with higher scores indicating a more preserved cognition.
Neuropsychiatric Inventory (NPI) | Change from baseline to week 2 and 12
  Neuropsychiatric Inventory (NPI) is designed to be a structured clinical interview about neuropsychiatric and behavioral symptoms will be assessed by; the score ranges from 0 (no symptoms) to 144 (severe symptoms).
Qualitive Pentagon Test | Change from baseline to week 2 and 12
  Praxis-constructive abilities will be assessed by Qualitive Pentagon Test; the subject is asked to copy two intersecting pentagons. Qualitive Pentagon Test scores range from 0 to 13, with higher scores indicating a better performance.
Rey Auditory Verbal Learning Test (RAVLT) | Change from baseline to week 2 and 12
  Verbal memory will be assessed using the Rey Auditory Verbal Learning Test (RAVLT), including immediate recall (sum of trials), delayed recall after 15 minutes. Scores reflect the number of correctly recalled items.
Trail Making Test (TMT - AB) | Change from baseline to week 2 and 12
  Executive function will be assessed using the Trail Making Test, including Part A (visual attention and processing speed) and Part B (task switching and cognitive flexibility). Higher completion times reflect poorer performance.
Clock Drawing Test (CDT) | Change from baseline to week 2 and 12
  Constructional praxis abilities, mental representation skills, and visuospatial planning will be evaluated by Clock Drawing Test (CDT). CDT scores range from 0 to 15, with higher scores indicating a better performance.
Rey-Osterrieth Complex Figure Test (ROCF) | Change from baseline to week 2 and 12
  Visuoconstructive abilities and visual memory will be assessed by Rey-Osterrieth Complex Figure. It requires the subject to copy a complex geometric figure and subsequently reproduce it from meory after a 10 minutes delay. Both tests score from 0 to 36, with higher score indicating a better performance.
Phonemic Fluency Test | Change from baseline to week 2 and 12
  Cognitive flexibility and verbal fluency will be evalueted by Phonemic Fluency Test. Subject is asked to generate as many words as possible from a given letter within a limited time (60 seconds); higher scores indicate better perfomance.
Semantic Fluency Test | Change from baseline to week 2 and 12
  Lexical-semantic access and executive functioning will be evalueted by Semantic Fluency Test. Subject is asked to generate as many words as possible from a given category within a limited time (60 seconds); higher scores indicate better perfomance.
Digit Span Test | Change from baseline to week 2 and 12
  Short-term memory and working memory will be assessed respectively using the Digit Span forward and Digit Span backward. Scores reflect the maximum number of digits recalled in correct order.
Visual Search Task | Change from baseline to week 2 and 12
  Attention and cognitive flexibility will be assessed using a Visual Search task. Participants will be instructed to identify and select a predefined target each time it appears on the screen. Performance will be quantified by the number of correct detections (hits), missed targets (omissions), and incorrect responses (errors).

SECONDARY OUTCOMES:
Change in Biological Markers | Change from baseline to week 2 and 12
  A venous blood draw (35 ml) will be performed at each timepoint (T0, T02, T12). The samples will be processed for serum, plasma, and DNA extraction. Neurodegeneration biomarkers will be analyzed, specifically changes in plasma neurofilament light (NfL) levels (pg/mL) will be evaluated. The plasma biomarker profile will be evaluated as a predictor of treatment efficacy and correlated with differential treatment response.
Change in electroencephalography (EEG) | Change from baseline to week 2 and 12
  Using resting-state electroencephalography (EEG) recorded under eyes-open and eyes-closed conditions, the investigators will assess changes in EEG alpha-band power (8-12 Hz). Alpha power will be quantified from scalp EEG recordings using spectral power analysis performed on the pre-processed EEG data.
Change in TMS-EEG | Change from baseline to week 2 and 12
  Cortical reactivity and effective connectivity will be assessed by analyzing TMS-evoked potentials, obtained from TMS-EEG coregistration after occipital cortex stimulation.
Basic Activities of Daily Living (BADL) | Baseline
  Basic Activities of Daily Living (BADL; range 0-6, higher scores indicating worse outcome) assesses the loss of daily self-sufficiency.
  It will be evaluated as predictors of treatment efficacy and examined for associations with differential treatment response.
Instrumental Activities of Daily Living (IADL) | Baseline
  Instrumental Activities of Daily Living (IADL; range 0-8, higher scores indicating worse outcome) assesses the loss of complex instrumental acitivities.
  It will be evaluated as predictors of treatment efficacy and examined for associations with differential treatment response.
Unified Parkinson's Disease Rating Scale - Part III (UPDRS-III) | Baseline
  Unified Parkinson's Disease Rating Scale - Part III (UPDRS-III; range 0-132, higher scores indicating worse outcome) assesses motor impairment.
  It will be evaluated as predictors of treatment efficacy and examined for associations with differential treatment response.
Demographic characteristics | Baseline
  Demographic characteristics (age, gender, and level of education) will be evaluated as predictors of treatment efficacy and examined for associations with differential treatment response.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Centro San Giovanni Di Dio - Fatebenefratelli Brescia, Brescia, Italy, Italy

REFERENCES:
- [Background] Aoki Y, Kazui H, Pascal-Marqui RD, Ishii R, Yoshiyama K, Kanemoto H, Suzuki Y, Sato S, Hata M, Canuet L, Iwase M, Ikeda M. EEG Resting-State Networks in Dementia with Lewy Bodies Associated with Clinical Symptoms. Neuropsychobiology. 2019;77(4):206-218. doi: 10.1159/000495620. Epub 2019 Jan 17. PMID 30654367
- [Background] Antal A, Alekseichuk I, Bikson M, Brockmoller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Floel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID 28709880
- [Background] Amodio P, Wenin H, Del Piccolo F, Mapelli D, Montagnese S, Pellegrini A, Musto C, Gatta A, Umilta C. Variability of trail making test, symbol digit test and line trait test in normal people. A normative study taking into account age-dependent decline and sociobiological variables. Aging Clin Exp Res. 2002 Apr;14(2):117-31. doi: 10.1007/BF03324425. PMID 12092785
- [Background] Bagattini C, Mutanen TP, Fracassi C, Manenti R, Cotelli M, Ilmoniemi RJ, Miniussi C, Bortoletto M. Predicting Alzheimer's disease severity by means of TMS-EEG coregistration. Neurobiol Aging. 2019 Aug;80:38-45. doi: 10.1016/j.neurobiolaging.2019.04.008. Epub 2019 Apr 13. PMID 31077959
- [Background] Benussi A, Cantoni V, Rivolta J, Zoppi N, Cotelli MS, Bianchi M, Cotelli M, Borroni B. Alpha tACS Improves Cognition and Modulates Neurotransmission in Dementia with Lewy Bodies. Mov Disord. 2024 Nov;39(11):1993-2003. doi: 10.1002/mds.29969. Epub 2024 Aug 13. PMID 39136447
- [Background] Bonato C, Miniussi C, Rossini PM. Transcranial magnetic stimulation and cortical evoked potentials: a TMS/EEG co-registration study. Clin Neurophysiol. 2006 Aug;117(8):1699-707. doi: 10.1016/j.clinph.2006.05.006. Epub 2006 Jun 22. PMID 16797232
- [Background] Bortoletto M, Veniero D, Thut G, Miniussi C. The contribution of TMS-EEG coregistration in the exploration of the human cortical connectome. Neurosci Biobehav Rev. 2015 Feb;49:114-24. doi: 10.1016/j.neubiorev.2014.12.014. Epub 2014 Dec 22. PMID 25541459
- [Background] Hoy KE, Bailey N, Arnold S, Windsor K, John J, Daskalakis ZJ, Fitzgerald PB. The effect of gamma-tACS on working memory performance in healthy controls. Brain Cogn. 2015 Dec;101:51-6. doi: 10.1016/j.bandc.2015.11.002. Epub 2015 Nov 12. PMID 26580743
- [Background] Massimini M, Ferrarelli F, Huber R, Esser SK, Singh H, Tononi G. Breakdown of cortical effective connectivity during sleep. Science. 2005 Sep 30;309(5744):2228-32. doi: 10.1126/science.1117256. PMID 16195466
- [Background] Monaco M, Costa A, Caltagirone C, Carlesimo GA. Forward and backward span for verbal and visuo-spatial data: standardization and normative data from an Italian adult population. Neurol Sci. 2013 May;34(5):749-54. doi: 10.1007/s10072-012-1130-x. Epub 2012 Jun 12. PMID 22689311
- [Background] Morishima Y, Akaishi R, Yamada Y, Okuda J, Toma K, Sakai K. Task-specific signal transmission from prefrontal cortex in visual selective attention. Nat Neurosci. 2009 Jan;12(1):85-91. doi: 10.1038/nn.2237. Epub 2008 Dec 21. PMID 19098905
- [Background] Morrin H, Fang T, Servant D, Aarsland D, Rajkumar AP. Systematic review of the efficacy of non-pharmacological interventions in people with Lewy body dementia. Int Psychogeriatr. 2018 Mar;30(3):395-407. doi: 10.1017/S1041610217002010. Epub 2017 Oct 9. PMID 28988547
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Treisman AM, Gelade G. A feature-integration theory of attention. Cogn Psychol. 1980 Jan;12(1):97-136. doi: 10.1016/0010-0285(80)90005-5. No abstract available. PMID 7351125
- [Background] Ragazzoni A, Pirulli C, Veniero D, Feurra M, Cincotta M, Giovannelli F, Chiaramonti R, Lino M, Rossi S, Miniussi C. Vegetative versus minimally conscious states: a study using TMS-EEG, sensory and event-related potentials. PLoS One. 2013;8(2):e57069. doi: 10.1371/journal.pone.0057069. Epub 2013 Feb 27. PMID 23460826
- [Background] McKeith IG, Boeve BF, Dickson DW, Halliday G, Taylor JP, Weintraub D, Aarsland D, Galvin J, Attems J, Ballard CG, Bayston A, Beach TG, Blanc F, Bohnen N, Bonanni L, Bras J, Brundin P, Burn D, Chen-Plotkin A, Duda JE, El-Agnaf O, Feldman H, Ferman TJ, Ffytche D, Fujishiro H, Galasko D, Goldman JG, Gomperts SN, Graff-Radford NR, Honig LS, Iranzo A, Kantarci K, Kaufer D, Kukull W, Lee VMY, Leverenz JB, Lewis S, Lippa C, Lunde A, Masellis M, Masliah E, McLean P, Mollenhauer B, Montine TJ, Moreno E, Mori E, Murray M, O'Brien JT, Orimo S, Postuma RB, Ramaswamy S, Ross OA, Salmon DP, Singleton A, Taylor A, Thomas A, Tiraboschi P, Toledo JB, Trojanowski JQ, Tsuang D, Walker Z, Yamada M, Kosaka K. Diagnosis and management of dementia with Lewy bodies: Fourth consensus report of the DLB Consortium. Neurology. 2017 Jul 4;89(1):88-100. doi: 10.1212/WNL.0000000000004058. Epub 2017 Jun 7. PMID 28592453
- [Background] Kujirai T, Caramia MD, Rothwell JC, Day BL, Thompson PD, Ferbert A, Wroe S, Asselman P, Marsden CD. Corticocortical inhibition in human motor cortex. J Physiol. 1993 Nov;471:501-19. doi: 10.1113/jphysiol.1993.sp019912. PMID 8120818
- [Background] Herrmann CS, Rach S, Neuling T, Struber D. Transcranial alternating current stimulation: a review of the underlying mechanisms and modulation of cognitive processes. Front Hum Neurosci. 2013 Jun 14;7:279. doi: 10.3389/fnhum.2013.00279. eCollection 2013. PMID 23785325
- [Background] Ferrarelli F, Massimini M, Peterson MJ, Riedner BA, Lazar M, Murphy MJ, Huber R, Rosanova M, Alexander AL, Kalin N, Tononi G. Reduced evoked gamma oscillations in the frontal cortex in schizophrenia patients: a TMS/EEG study. Am J Psychiatry. 2008 Aug;165(8):996-1005. doi: 10.1176/appi.ajp.2008.07111733. Epub 2008 May 15. PMID 18483133
- [Background] Cromarty RA, Elder GJ, Graziadio S, Baker M, Bonanni L, Onofrj M, O'Brien JT, Taylor JP. Neurophysiological biomarkers for Lewy body dementias. Clin Neurophysiol. 2016 Jan;127(1):349-359. doi: 10.1016/j.clinph.2015.06.020. Epub 2015 Jun 27. PMID 26183755
- [Background] Costa A, Bagoj E, Monaco M, Zabberoni S, De Rosa S, Papantonio AM, Mundi C, Caltagirone C, Carlesimo GA. Standardization and normative data obtained in the Italian population for a new verbal fluency instrument, the phonemic/semantic alternate fluency test. Neurol Sci. 2014 Mar;35(3):365-72. doi: 10.1007/s10072-013-1520-8. Epub 2013 Aug 21. PMID 23963806
- [Background] Caffarra P, Gardini S, Zonato F, Concari L, Dieci F, Copelli S, Freedman M, Stracciari A, Venneri A. Italian norms for the Freedman version of the Clock Drawing Test. J Clin Exp Neuropsychol. 2011 Nov;33(9):982-8. doi: 10.1080/13803395.2011.589373. Epub 2011 Aug 1. PMID 22082081
- [Background] Caffarra P, Vezzadini G, Dieci F, Zonato F, Venneri A. Rey-Osterrieth complex figure: normative values in an Italian population sample. Neurol Sci. 2002 Mar;22(6):443-7. doi: 10.1007/s100720200003. PMID 11976975
- [Background] Carlesimo GA, De Risi M, Monaco M, Costa A, Fadda L, Picardi A, Di Gennaro G, Caltagirone C, Grammaldo L. Normative data for measuring performance change on parallel forms of a 15-word list recall test. Neurol Sci. 2014 May;35(5):663-8. doi: 10.1007/s10072-013-1573-8. Epub 2013 Nov 12. PMID 24218156
- [Background] Chatzikonstantinou S, McKenna J, Karantali E, Petridis F, Kazis D, Mavroudis I. Electroencephalogram in dementia with Lewy bodies: a systematic review. Aging Clin Exp Res. 2021 May;33(5):1197-1208. doi: 10.1007/s40520-020-01576-2. Epub 2020 May 7. PMID 32383032